CLINICAL TRIAL: NCT01359332
Title: Evaluation of the Interests of a Therapeutic Hypothermia Procedure in Convulsive Status EPILEPTICUS in Adults in Intensive Care - HYBERNATUS Study
Brief Title: Evaluation of Therapeutic Hypothermia in Convulsive Status EPILEPTICUS in Adults in Intensive Care
Acronym: HYBERNATUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081249
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Convulsive Status EPILEPTICUS
Keywords: Convulsive status EPILEPTICUS; hypothermia therapy; (defined as continuous SEIZURING for longer than 5 min or three seizures; not separated by recovery of normal consciousness; or of the level of consciousness present before the; seizures)
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypothermia (Experimental)
  Interventions: Procedure: Moderate hypothermia
- control (No Intervention)

INTERVENTIONS:
Procedure: Moderate hypothermia — procedure of moderate hypothermia therapy, between 32 ° and 34 ° C for 24 hours
  Arms: hypothermia

SUMMARY:
Status EPILEPTICUS (SE) is a major medical emergency. The incidence per 100,000 population has been estimated at 9.9 episodes in Europe and 41 episodes in the US. The overall morbidity and mortality associated with convulsive SE (CSE) is 60% at three months. The alteration of functional prognosis of these patients is more conventionally attributed to the cause than to CSE itself. Longer seizure duration, progression to refractory status EPILEPTICUS and presence of cerebral insult are strong factors independently associated with a poor functional outcome. These three factors offer may be amenable to improvement and hope for preventive strategies. Current guidelines recommend the use of anticonvulsant treatment whose goal is prompt cessation of clinical and electrical seizures. None of these treatments has demonstrated NEUROPROTECTICE property. Therapeutic moderate hypothermia (between 32 and 34 ° C) showed interest in neuroprotection of post anoxic coma patients after a cardiovascular arrest on ventricular fibrillation by reducing morbidity and mortality in about 20% without major side effects. This technique has been used successfully in various pathologies such as stroke or traumatic brain injury. Pathophysiological mechanisms involved in epileptogenesis and neurotoxicity induced by persistence of seizures can be blocked by therapeutic hypothermia. Recent work on experimental models of SE demonstrated neuroprotective and anticonvulsant interest of therapeutic hypothermia. Therapeutic hypothermia has also been successfully used in some cases of particularly refractory CSE. Its early use in patients with SE would have a double interest: neuroprotective and anticonvulsant. There is currently no published studies or ongoing to determine the interest of its early use in patients with CSE.

DETAILED DESCRIPTION:
Status EPILEPTICUS (SE) is a major medical emergency. The incidence per 100,000 population has been estimated at 9.9 episodes in Europe and 41 episodes in the US. The overall morbidity and mortality associated with convulsive SE (CSE) is 60% at three months. The alteration of functional prognosis of these patients is more conventionally attributed to the cause than to CSE itself. Longer seizure duration, progression to refractory status EPILEPTICUS and presence of cerebral insult are strong factors independently associated with a poor functional outcome. These three factors offer may be amenable to improvement and hope for preventive strategies. Current guidelines recommend the use of anticonvulsant treatment whose goal is prompt cessation of clinical and electrical seizures. None of these treatments has demonstrated NEUROPROTECTICE property. Therapeutic moderate hypothermia (between 32 and 34 ° C) showed interest in neuroprotection of post anoxic coma patients after a cardiovascular arrest on ventricular fibrillation by reducing morbidity and mortality in about 20% without major side effects. This technique has been used successfully in various pathologies such as stroke or traumatic brain injury. Pathophysiological mechanisms involved in epileptogenesis and neurotoxicity induced by persistence of seizures can be blocked by therapeutic hypothermia. Recent work on experimental models of SE demonstrated neuroprotective and anticonvulsant interest of therapeutic hypothermia. Therapeutic hypothermia has also been successfully used in some cases of particularly refractory CSE. Its early use in patients with SE would have a double interest: neuroprotective and anticonvulsant. There is currently no published studies or ongoing to determine the interest of its early use in patients with CSE.

Thus, the current study AIMAS at evaluating the effectiveness of the implementation of a procedure of moderate hypothermia therapy, between 32 ° and 34 ° C for 24 hours, to reduce morbidity and mortality at 3 months (+ / - 1 week) in mechanically ventilated ICU patients with convulsive status EPILEPTICUS.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥ 18 years
* patient hospitalized in intensive care unit
* patient already under mechanical ventilation
* patient who presented a convulsive status EPILEPTICUS episode (defined as continuous SEIZURING for longer than 5 min or three seizures not separated by recovery of normal consciousness or of the level of consciousness present before the seizures)
* whose motor manifestations had begun less than 8 hours before randomization
* after having informed written consent signed by a parent or a close if present.

Exclusion Criteria:

* patients with full recovery, postanoxic status EPILEPTICUS after cardia arrest
* convulsive status EPILEPTICUS for which an intervention (neurosurgical or other) is urgently needed not allowing the application of the procedure for therapeutic hypothermia
* dying patient, limitations in care, or whose life expectancy is estimated at baseline of less than 1 year
* patients whose follow-up to 3 months (+ / - 1 week) seems a PRIORI not possible
* pregnant women (pregnancy positive urine test or known before inclusion),
* participation in another biomedical therapeutic intervention whose primary endpoint was not reached at inclusion in HYBERNATUS study
* not affiliation to a social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Functional impairment at 3 months | 3 months
  Functional impairment is defined by a Glasgow Outcome Scale strictly less than 5.
  The time of evaluation should be 3 months (+/- 1 week)

SECONDARY OUTCOMES:
mortality | hospital discharge
mortality | ICU discharge
mortality | 90 days
Incidence of functional sequelae | 3 months
  Judged on the frequency of seizures, the recurrence of epileptic status after hospitalization, the number of anti-epileptic drug, mini mental score (MMS).
length of icu stay | 3 months
length of hospital stay | 3 months
Percentages of convulsive and non-convulsive seizure recurrences | 6 to 12 hours
  Progression to status epilepticus
Seizure duration in minutes | 3 days
Percentage of refractory status epilepticus cases | 3 days
  Judged on the frequency of seizures within 24 hours after status epilepticus onset (refractory status epilepticus on day 1) and on the frequency of seizures within 48 hours after anesthetic treatment withdrawal (super refractory status epilepticus)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane LEGRIEL, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital André MIGNOT- Service de réanimation médico-chirurgical, Le Chesnay, France

REFERENCES:
- [Derived] Jacq G, Crepon B, Resche-Rigon M, Schenck M, Geeraerts T, Meziani F, Megarbane B, Chaffaut C, Cariou A, Legriel S. Clinician-Reported Physical and Cognitive Impairments After Convulsive Status Epilepticus: Post Hoc Study of a Randomized Controlled Trial. Neurocrit Care. 2024 Apr;40(2):495-505. doi: 10.1007/s12028-023-01758-6. Epub 2023 Jun 7. PMID 37286846
- [Derived] Fontaine C, Lemiale V, Resche-Rigon M, Schenck M, Chelly J, Geeraerts T, Hamdi A, Guitton C, Meziani F, Lefrant JY, Megarbane B, Mentec H, Chaffaut C, Cariou A, Legriel S; HYBERNATUS Study Group. Association of systemic secondary brain insults and outcome in patients with convulsive status epilepticus: A post hoc study of a randomized controlled trial. Neurology. 2020 Nov 3;95(18):e2529-e2541. doi: 10.1212/WNL.0000000000010726. Epub 2020 Sep 10. PMID 32913029
- [Derived] Legriel S, Lemiale V, Schenck M, Chelly J, Laurent V, Daviaud F, Srairi M, Hamdi A, Geri G, Rossignol T, Hilly-Ginoux J, Boisrame-Helms J, Louart B, Malissin I, Mongardon N, Planquette B, Thirion M, Merceron S, Canet E, Pico F, Tran-Dinh YR, Bedos JP, Azoulay E, Resche-Rigon M, Cariou A; HYBERNATUS Study Group. Hypothermia for Neuroprotection in Convulsive Status Epilepticus. N Engl J Med. 2016 Dec 22;375(25):2457-2467. doi: 10.1056/NEJMoa1608193. PMID 28002714
- [Derived] Legriel S, Pico F, Tran-Dinh YR, Lemiale V, Bedos JP, Resche-Rigon M, Cariou A. Neuroprotective effect of therapeutic hypothermia versus standard care alone after convulsive status epilepticus: protocol of the multicentre randomised controlled trial HYBERNATUS. Ann Intensive Care. 2016 Dec;6(1):54. doi: 10.1186/s13613-016-0159-z. Epub 2016 Jun 21. PMID 27325409